CLINICAL TRIAL: NCT07106281
Title: Effect of Chronic Grape Extract Supplementation in Trained Cross-training Athletes: A Randomized, Triple-blinded, Placebo-Controlled Crossover Study
Brief Title: Chronic Grape Extract in Crosstraining Athletes: A Randomized Crossover Trial
Acronym: CROSSUVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Universidad de La Laguna, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain. (Unknown)
Responsible Party: Principal Investigator, Lucas Jurado-Fasoli, PhD, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CROSSUVA
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Performance
Keywords: grape seed extract; muscle damage; concurrent exercise; nutrition; recovery
MeSH Terms: interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grape seed extract (Experimental): 600 mg of Grape seed extract
  Interventions: Dietary Supplement: Grape Seed Extract
- Placebo (Placebo Comparator): Preparation of colorants, sweeteners, aromas, and acidulants
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Grape Seed Extract — 600mg of Grape Seed Extract
  Arms: Grape seed extract
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effect of cronic GSE intake in crosstraining may have a favorable impact on biochemical markers, recovery, and performance.

DETAILED DESCRIPTION:
Supplementation with certain antioxidant nutrients is a feasible strategy to accelerate recovery from fatigue and prevent exercise-induced oxidative damage. Grape seed extract (GSE) contains flavonoids such as proanthocyanidins, which are potent antioxidants with numerous health benefits. Therefore, optimizing the recovery process after training is essential for athletes engaged in strength and power sports who aim to enhance performance.

Thirty trained CrossFit athletes consumed grape seed extract or a placebo for one week. The training session consisted of a 12-minute strength block, a 13-minute metabolic conditioning (MetCon), and a final 15-minute MetCon. The Rating of Perceived Exertion (RPE), Gastrointestinal Distress Score (GDS), blood pressure and the Perceived Recovery Status scale (RPS) were administered at the beginning of the session and at the end of each segment of the CrossFit session. DOMS was assessed using a visual analog scale at 24 and 48 hours after the CrossFit session.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years.
* Body mass index: 18.5-30 kg/m2.
* Ability to understand the instructions, objectives, and study protocol.
* Minimum of 3 years of experience in crosstraining, with at least 6 hours of weekly training over the past 3 months.
* Resident on the island of Tenerife.

Exclusion Criteria:

* History of a significant adverse cardiovascular event, renal insufficiency, cirrhosis, eating disorder, weight control surgical intervention, or type 2 diabetes mellitus.
* Any chronic pathology in which the intake of nutritional supplements, especially use of antioxidant supplements during the 4 weeks prior to the start of the study.
* Any condition that, in the investigator's judgment, would impair the ability to participate in the study or represent a personal risk to the participant.
* Use of medications that may affect the study results.
* Unstable body weight for 3 months prior to the start of the study (> 4 kg loss or gain in weight).
* Active tobacco abuse or illicit drug use, or history of treatment for alcohol abuse.
* On a special diet or prescribed for other reasons (e.g., celiac disease).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Performance | 48 hours
  Performance measured through the countermovement jump
Performance | 60 minutes
  Deep squat test at 70% of repetition maximum

SECONDARY OUTCOMES:
Attention | 60 minutes
  Selective attention and inhibitory control measured by the Stroop test
Performance: Weight used in the crosstraining session | 60 minutes
  Weight used in the crosstraining session
Performance: Time performed in the crosstraining session | 60 minutes
  Time performed in the crosstraining session
Subjective fatigue throug the the RPE scale | 60 minutes
  Rate of perceived exertion scale
Gastrointestinal distress | 60 minutes
  Gastrointestinal distress through the Gastrointestinal Distress Score (GDS)
Recovery | 60 minutes
  Perceived Recovery Status Scale (RPS)
Delayed-onset muscle soreness (DOMS) | 24 hours
  Delayed-onset muscle soreness (DOMS) scale (0-10 arbitrary units)
Capillar lactate levels | 60 minutes
  Capillar lactate levels
Heart rate | 60 minutes
  Heart rate
Blood pressure | 60 minutes
  Blood pressure
Biochemical parameters | 48 hours
  Biochemical parameters of muscle damage: Glutamate oxaloacetate transaminase (GOT), glutamate pyruvate transaminase (GPT), creatine kinase (CK), urea, lactate dehydrogenase (LDH), myoglobin, glutathione peroxidase (GPx), catalase, superoxide dismutase (SOD), and interleukin 6 (IL-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de la Laguna, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided